CLINICAL TRIAL: NCT07216183
Title: Epidermal Sensors for Wireless and Enhanced Amputee Skin Tracking (E-SWEAT) Part 1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Amay Bandodkar, Assistant Professor, North Carolina State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 26923; HT9425-24-1-0579 (Other Grant/Funding Number: Department of Defense, U.S.)
Record Dates: First submitted 2025-09-11; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Transtibial Amputation
Keywords: sweat biomarker; prosthetic socket; pressure ulcer; residual limb health
MeSH Terms: conditions — Pressure Ulcer | interventions — Walking

STUDY DESIGN:
Intervention Model Description: The participants are exposed to the two tasks in randomly decided sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Normal walking (Experimental): Participants walk on a treadmill with user preferred speed.
  Interventions: Procedure: Walk; Device: E-SWEAT Sensor
- No load excise - Yuga post (Active Comparator): Participants conduct a yuga post which involves their efforts but not load on their residual limbs
  Interventions: Procedure: Yuga post; Device: E-SWEAT Sensor

INTERVENTIONS:
Procedure: Walk — Treadmill walking
  Arms: Normal walking
Procedure: Yuga post — Participants conduct a yuga post which involves their efforts but not load on their residual limbs
  Arms: No load excise - Yuga post
Device: E-SWEAT Sensor — Mounting the E_SWEAT sensor to monitor the lactic density, pressure, and temperature inside the socket

SUMMARY:
The goal of this clinical trial is to 1) demonstrate the feasibility of monitoring pressure, temperature, and lactic acid density of sweat inside the prosthetic socket, and 2) verify the relationship between mechanical pressure and Lactic acid density of sweat for lower limb amputees among transtibial amputees. The main questions it aims to answer are:

* Is it feasible to reliably monitor pressure, temperature, and lactic acid density inside the prosthetic sockets simultaneously?
* Will the lactic acid density increase with higher pressure exposure? The participants are expected to wear the newly developed E-SWEAT system on their residual limb and are exposed to two activities, walk which generate mechanical load on the residual limb, and a yoga post - birddog, which does not generate mechanical loading on the residual limb. The E-SWEAT will measure pressure, temperature, and lactic acid density of sweat during these tasks.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Have a unilateral lower limb amputee (below the knee). The tibial length on the residual limb must be greater than half of the length of the tibial on the unaffected side
* Have an amputation that occurred over 2 years ago
* Have at least 1 year of experience using your prosthetic leg
* Have used the current socket for at least 6 months without a significant skin issue or major modification
* Be able to comfortably walk 6 mins (with prosthetic legs) without pausing to rest
* Be willing to come to North Carolina State University's Centennial Campus to participate in research and be photographed while doing research activities

Exclusion Criteria:

* Have a cognitive or visual impairment that affects the participant's ability to provide informed consent or to follow simple instructions during the experiments
* Have any neuropathy observed on the residual limb
* Experience numbness, tingling, muscle weakness, and/or pain in your residual limb
* Weigh more than 300lbs
* Do not want to take photos
* Are pregnant or plan to get pregnant
* Are allergic to latex, which is often contained in medical tapes.
* If you are using medication to control sweat on your residual limb, and your medical provider does not think that it is OK to avoid these medications for 48 hours.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Lactic acid density | periprocedural in the first visit
  amount of lactic acid in sweat

SECONDARY OUTCOMES:
Socket environment - temperature | periprocedural in the first visit
  temperature at the location where the E-SWEAT is mounted
Socket environment - pressure | periprocedural in the first visit
  Pressure measured at the location where the E-SWAET is mounted

OTHER OUTCOMES:
Body weight | At the beginning of the first visit
  Participants' body weight

CONTACTS AND LOCATIONS:
Locations (1):
- Engineering Build III, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All data will be coded with an ID, which randomly generated.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT07216183/ICF_000.pdf